CLINICAL TRIAL: NCT03438318
Title: A Multicenter, Two-Part, Phase 1B Clinical Study of CMP-001 in Combination With Atezolizumab With and Without Radiation Therapy in Subjects With Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: Study Evaluating CMP-001 in Combination With Atezolizumab in Participants With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-003
Record Dates: First submitted 2018-01-25; First posted 2018-02-19 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (CMP-001, Atezolizumab and Optional Radiation Therapy) (Experimental): Participants will receive CMP-001 5 milligrams (mg) SC once weekly for 2 weeks, then 10 mg IT once weekly for 3 weeks, followed by every 3 weeks thereafter until discontinuation of treatment in combination with atezolizumab SC every 3 weeks starting at Week 2. Route of administration (IT/SC) for CMP-001 beyond Week 5 will be determined by Investigator. Participants enrolled in Part A who progressed per RECIST v1.1 on combination of CMP-001 and atezolizumab have opportunity to enroll in Part A optional radiation therapy add-on after documented disease progression per CT/MRI or PET scan. After CMP-001 washout period of 10 days, participants will be treated with radiation consisting of 20 grays in 5 fractions for 5 days then resume CMP-001 treatment.
  Interventions: Drug: CMP-001; Drug: Atezolizumab; Radiation: Radiation Therapy
- Part B (Radiation Therapy, CMP-001 and Atezolizumab) (Experimental): Participants will be treated with radiation therapy consisting of 20 grays in 5 fractions for 5 days, then participants will receive CMP-001 5 mg SC once weekly for 2 weeks, then 10 mg IT once weekly for 3 weeks, followed by dosing every 3 weeks thereafter until discontinuation of treatment. The route of administration (that is, IT or SC) for CMP-001 beyond Week 5 will be determined by the Investigator. First dose of CMP-001 will be administered within 2 days of radiation therapy. Atezolizumab will be administered SC in combination with CMP-001 every 3 weeks starting at Week 2.
  Interventions: Drug: CMP-001; Drug: Atezolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: CMP-001 — CMP-001 will be administered as per the dose and schedule specified in the respective arms.
Drug: Atezolizumab — Atezolizumab will be administered as per the approved label and according to the schedule specified in the respective arms.
Radiation: Radiation Therapy — Radiation therapy will be administered using either 3-dimensional (3D) conformal radiotherapy or intensity-modulated radiation therapy (IMRT) to non-target node or metastatic lesion as per the dose and schedule specified in the respective arms.

SUMMARY:
This is a multicenter, two part (Part A and Part B) clinical study of CMP-001 administered intratumorally (IT) and subcutaneously (SC) in combination with atezolizumab with or without radiation therapy in participants with NSCLC.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals

This study will be conducted in two parts, run sequentially: Part A of the study will evaluate the safety and preliminary signs of efficacy for the combination of CMP-001 and atezolizumab. Part B of the study will evaluate the addition of radiation therapy to the combination of CMP-001 and atezolizumab.

Each part of the study will follow a Simon 2-stage Optimal Design approach. Part A and Part B of the study will commence with a safety run in of 5 participants treated with the combination treatment (CMP-001 and atezolizumab in Part A; and CMP-001, atezolizumab and radiation therapy in Part B). After the first 5 participants have passed a safety dose-limiting toxicity (DLT) observation period of 30 days and upon approval from the Safety Review Committee (SRC), both parts of the study will continue with enrollment of an additional 7 participants in each part to complete Stage 1 of respective parts. If an acceptable safety profile is established and at least 2 responders out of 12 evaluable participants (that is, complete and partial responders based on Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 [v1.1] or RECIST v1.1 for immune-based therapeutics [iRECIST] criteria) in Stage 1), the study will enroll an additional 23 evaluable participants in Stage 2 of each part. A maximum of 35 evaluable participants will be enrolled in each Part A and Part B.

Participants enrolled in Part A with documented progression per RECIST v1.1 on the combination of CMP-001 and atezolizumab have the option to receive radiation therapy add-on treatment after documented disease progression per computed tomography (CT)/magnetic resonance imaging (MRI) or positron emission tomography (PET) scan. The total number of participants enrolled into the Part A optional radiation therapy add-on may not exceed the total number of participants enrolled in Part A. Enrollment of participants in Part A optional radiation therapy add-on will not affect enrollment in Part B of the study as these participants will be evaluated separately.

Participants will continue treatment with CMP-001 in combination with atezolizumab as long as they do not experience unacceptable toxicities and when, according to the Investigator, continued treatment is in the participant's best interest.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of metastatic NSCLC.
* Documented disease progression on prior programmed cell death-1/programmed death-ligand 1 (PD-1/PD-L1) therapy in any line. Participants must have received a minimum of 4 doses of anti-PD-1/PD-L1 therapy before enrolling into the CMP-001-003 study. If participants have received fewer than 4 doses of anti-PD-1/PD-L1 therapy, documented radiologic progression and sponsor approval is necessary prior to inclusion.
* Participants with epidermal growth factor (EGFR) activating mutations, EGFR T790M or anaplastic lymphoma kinase (ALK) gene re-arrangement must have received prior standard of care and have evidence of disease progression. With the exception of participants with squamous cell cancer, EGFR and ALK status must be known prior to enrollment.
* Participants must have at least one extra-central nervous system (CNS), non-bone tumor lesion amenable for IT injection greater than or equal to (>=) 1.5 centimeters (cm) and that is not in close proximity or encasing crucial structures such as major blood vessels, trachea, nerve bundles.
* Measurable disease per RECIST version 1.1.
* Capable of understanding and complying with protocol requirements.
* A life expectancy of greater than 24 weeks at Screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at Screening.
* Most recent laboratory values within 2 weeks prior to Week 1 Day 1 meet the following standards:

  1. Bone marrow function: Neutrophil count >=1,500/ cubic millimeters (mm^3) without granulocyte colony stimulating factor; Platelet count >=100,000/mm^3 without transfusion; Hemoglobin concentration >=9.0 grams per deciliter (g/dL).
  2. Liver function: Total bilirubin less than or equal to (<=) 2.0 times the upper limit of normal (ULN) of each institution with the exception of participants with Gilbert Disease serum bilirubin >= 3 * ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5 times the ULN with the following exceptions: participants with documented liver metastases; AST and ALT <=5 * ULN.
  3. Renal function: serum creatinine <=1.5 times the ULN.
  4. Lactate dehydrogenase (LDH) <=2 times ULN.
  5. Partial thromboplastin time (PTT) and international normalized ratio (INR): Activated PTT (aPTT) <=1.5 * ULN, unless related to lupus anticoagulant. Participants receiving unfractionated heparin must have aPTT between 1.5 and 2.5 * ULN or determined by their physician; INR < =1.5 * ULN. Participants receiving warfarin should have INR between 2.0 and 3.0 or within a range determined by their physician.
* The participant must sign a written informed consent form prior to the initiation of any study procedures. Adult participants unable to provide written informed consent on their own behalf will not be eligible for the study.
* For participants enrolled in Part B, metastatic lesions must be accessible for radiation therapy (that is, no direct overlap of the current treatment).

Exclusion Criteria:

* Pregnant or breastfeeding
* Received investigational therapy (that is, small molecule or biologic) within 30 days prior to the start of CMP-001 dosing on Week 1 Day 1. However, if an investigational therapy has a short half-life, a reduced wash out period may be acceptable with Sponsor approval. Acceptable washout periods for non-investigational therapy include:

  1. 3-14 days from prior tyrosine kinase inhibitor (TKI) depending on half-life.
  2. 3 weeks from prior chemotherapy.
  3. 1 week for prior palliative radiation therapy, or 2 weeks if prior brain radiation therapy.
  4. Received treatment with anti- cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody within 30 days prior to the start of CMP-001.
  5. 14 days for prior PD-1 therapy.
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). If there is no known or documented history of HIV, HBV or HCV, the site is not required to do additional testing for these values at Screening.
* Developed autoimmune disorders of Grade 4 while on prior immunotherapy. Participants who developed autoimmune disorders, of Grade <=3 may enroll if the disorder has resolved to Grade <=1 and the participant has been off systemic steroids at doses greater than (>) 10 milligrams per day (mg/day), for the treatment of the autoimmune disorder, for at least 2 weeks.
* Require systemic pharmacologic doses of corticosteroids greater than the equivalent of 10 mg/day prednisone; topical, ophthalmologic and inhalational steroids are permitted. Participants who have a history of adrenal insufficiency and are receiving greater than 10 mg/day prednisone may be eligible but only after Sponsor consultations. Participants who are currently receiving steroids at a dose of <=10 mg/day do not need to discontinue steroids prior to enrollment.
* Active (that is, symptomatic or progressing) CNS metastases. However, participants with active CNS metastases are eligible for the trial if:

  1. The metastases have been treated by surgery and/or radiotherapy.
  2. The participant is off corticosteroids of >10 mg/day prednisone or equivalent.
  3. The participant is neurologically stable for at least 2 weeks prior to Screening.
  4. Brain MRI completed within 6 weeks of Screening (required for all participants).
* Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator, would make the participant unable to cooperate or participate in the trial.
* Severe uncontrolled cardiac disease within 6 months of screening, including but not limited to uncontrolled hypertension; unstable angina; myocardial infarction (MI) or cerebrovascular accident (CVA).
* Requires prohibited treatment (that is., non-protocol specified anticancer pharmacotherapy, surgery or conventional radiotherapy for treatment of malignant tumor). Limited field single dose radiotherapy for pain palliation would be allowed at any time during the course of treatment.
* Women of childbearing potential who are unable or unwilling to use an acceptable method of contraception.
* Requires continuous anti-coagulation or anti-platelet therapy that cannot be safely interrupted to allow for IT injection and/or history of coagulopathy.
* History of another malignancy except for:

  1. Malignancy treated with curative intent and with no known active disease >5 years prior to the start of CMP-001 dosing on Week 1 Day 1 and of low potential risk for recurrence.
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  3. Adequately treated carcinoma in situ without evidence of disease (for example, cervical cancer in situ), superficial bladder cancer, squamous cell carcinoma of the skin, basal cell carcinoma of the skin.
  4. Other concurrent low-grade malignancies such as chronic lymphocytic leukemia (CLL) (Rai 0) may be considered after discussion and permission from Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Part A and B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of CMP-001 (Week 1 Day 1) until 30 days after the last CMP-001 injection (up to approximately 2 years 9 months)
  TEAEs will be evaluated and assigned a grade using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Part A and B: DLT | First 30 days of therapy starting from Week 1 Day 1

SECONDARY OUTCOMES:
Part A and B: Oral Temperature | From screening up to end of treatment (EOT) (up to approximately 2 years 9 months)
  Oral temperature should be measured in supine or seated position, following at least 3 minutes of rest.
Part A and B: Respiratory Rate | From screening up to EOT (up to approximately 2 years 9 months)
  Respiratory rate should be measured in supine or seated position, following at least 3 minutes of rest.
Part A and B: Systolic and Diastolic Blood Pressure | From screening up to EOT (up to approximately 2 years 9 months)
  Blood pressure should be measured in supine or seated position, following at least 3 minutes of rest.
Part A and B: Body Weight | From screening up to EOT (up to approximately 2 years 9 months)
  Physical examination included body weight measurement.
Part A and B: Body Mass Index (BMI) | From screening up to EOT (up to approximately 2 years 9 months)
  Physical examination included BMI measurement.
Part A and B: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG) Parameters | From screening up to EOT (up to approximately 2 years 9 months)
  ECG parameters will include heart rate and PR, QRS, QT, and QT corrected for heart rate (QTc) intervals. QT will be corrected using Fridericia's (QTcF) formula. ECG will be performed after the participant has been resting in supine or semi-supine position for at least 5 minutes.
Part A and B: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters | From screening up to EOT (up to approximately 2 years 9 months)
  Clinical laboratory parameters include serum chemistry, hematology, and urinalysis.
Part A and B: Concentration of Chemokine IP-10 | Day 1 of Weeks 1, 3, 8, and Day 2 of Weeks 3, 8
Part A and B: Objective Response Rate (ORR) (Percentage of Participants With Objective Response) as per RECIST V1.1 or iRECIST Using CT/PET or MRI Scans | Baseline until confirmed disease progression (CR or PR) or death, whichever occur first (assessment at every 9 weeks throughout the study from Week 1 Day 1, up to approximately 2 years 9 months
  ORR will be calculated as the number of participants with a confirmed complete response (CR) or partial response (PR) divided by the number of participants dosed.
Part A and B: Time to Response (TTR) as per RECIST V1.1 or iRECIST Using CT/PET or MRI Scans | From first dose of CMP-001 until disease progression or death, whichever occur first (assessment at every 9 weeks throughout the study from Week 1 Day 1, up to approximately 2 years 9 months)
Part A and B: Duration of Response (DOR) as per RECIST V1.1 or iRECIST Using CT/PET or MRI Scans | From the date of first confirmed CR or PR until the first date of recurrent or progressive disease (assessment at every 9 weeks throughout the study from Week 1 Day 1, up to approximately 2 years 9 months)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Medical Center, Duarte, California
  - University of Colorado Aurora, Aurora, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Negrao MV, Papadimitrakopoulou VA, Price AC, Tam AL, Furqan M, Laroia ST, Massarelli E, Pacheco J, Heymach JV, Tsao AS, Walker GV, Vora L, Mauro D, Kelley H, Wooldridge JE, Krieg AM, Niu J. Vidutolimod in Combination With Atezolizumab With and Without Radiation Therapy in Patients With Programmed Cell Death Protein 1 or Programmed Death-Ligand 1 Blockade-Resistant Advanced NSCLC. JTO Clin Res Rep. 2022 Oct 26;4(3):100423. doi: 10.1016/j.jtocrr.2022.100423. eCollection 2023 Mar. PMID 36925644